CLINICAL TRIAL: NCT01234324
Title: An Open Label Randomized Controlled Phase II Trial of Panitumumab in Combination With Epirubicin, Cisplatin and Capecitabine (ECX) Versus ECX Alone in Subjects With Locally Advanced Gastric Cancer or Cancer of the Gastroesophageal Junction.
Brief Title: ECX + Panitumumab vs. ECX Alone in Locally Advanced Gastric Cancer or Cancer of the Gastroesophageal Junction
Acronym: NEOPECX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Amgen (Industry); WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO/CAO-STO-0801; 2008-007798-18 (EudraCT Number)
Record Dates: First submitted 2010-10-28; First posted 2010-11-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Stomach Neoplasms; Gastroesophageal Junction Neoplasms
Keywords: Stomach Neoplasms; Gastroesophageal Junction Neoplasms; gastric cancer; cancer of the gastroesophageal junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Cisplatin; Capecitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: ECX + Panitumumab (Experimental)
  Interventions: Drug: Epirubicin, Cisplatin, Capecitabine, Panitumumab
- Arm 2: EXC alone (Active Comparator)
  Interventions: Drug: Epirubicin, Cisplatin, Capecitabine

INTERVENTIONS:
Drug: Epirubicin, Cisplatin, Capecitabine, Panitumumab — Epirubicin: 50mg/m², administered as an intravenous bolus over 10min on day 1 of each 21 day cycle; Cisplatin: 60mg/m², administered as an intravenous infusion over 4h on day 1 of each 21 day cycle; Capecitabine: 625mg/m², administered orally twice daily on each day of each 21 day cycle; Panitumumab: 9 mg/kg bodyweight, administered IV by an infusion pump through a peripheral line or catheter over 60 min +-15 min on day 1 of each 21 day cycle. Number of Cycles: 3 neoadjuvant cycles and 3 adjuvant cycles until disease progression, withdrawal of consent or unacceptable toxicity develops.
  Other Names: Xeloda®
  Arms: Arm 1: ECX + Panitumumab
Drug: Epirubicin, Cisplatin, Capecitabine — Epirubicin: 50mg/m², administered as an intravenous bolus over 10min on day 1 of each 21 day cycle; Cisplatin: 60mg/m², administered as an intravenous infusion over 4h on day 1 of each 21 day cycle; Capecitabine: 625mg/m², administered orally twice daily on each day of each 21 day cycle. Number of Cycles: 3 neoadjuvant cycles and 3 adjuvant cycles until disease progression, withdrawal of consent or unacceptable toxicity develops.
  Other Names: Vectibix®, Xeloda®
  Arms: Arm 2: EXC alone

SUMMARY:
That panitumumab in combination with Epirubicin, Cisplatin and Capecitabine (ECX) will safely decrease the frequency of pT3/T4 below that of ECX alone in subjects with locally advanced adenocarcinoma of the stomach and gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

* Competent to comprehend, sign, and date an IEC-approved informed consent form, written informed consent.
* Of either gender and aged 18 years or more.
* Diagnosed with histologically confirmed adenocarcinoma of the stomach or the gastroesophageal junction of Type I/II/III according to the classification of Siewert et al, 1996.
* Stage uT/3 or 4 N0/+ and M0 disease evaluated by endoscopic ultrasound, spiral computed tomography of the chest, abdomen and pelvis and by laparoscopy in uT3/T4 tumors.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Leucocyte count > 3,000/mm3.
* Platelet count ≥100,000/mm3.
* Haemoglobin ≥10 g/dl.
* Serum creatinine ≤ 1.5x of upper limit of normal (ULN).
* Creatinine clearance > 60 ml/kg/min measured either by 24-h urine sampling or calculated by using the Cockcroft-Gault formula .
* Aspartate aminotransferase (AST) ≤3 x ULN.
* Alanine aminotransferase (ALT) ≤3 x ULN.
* Bilirubin ≤ 1.5 x ULN.
* Magnesium ≥ lower limit of normal.
* Calcium ≥ lower limit of normal.
* Subject is deemed a good candidate for surgery.

Exclusion Criteria:

* Any metastatic disease.
* Other malignant tumours less than five years old. Exceptions include basocellular carcinoma, in situ cancer of the cervix of the uterus, or any curatively-treated other malignancies without evidence of disease for more than five years.
* Significant ascites or pleural effusion.
* Prior anti-EGFr antibody therapy (e.g. cetuximab) or treatment with small molecule EGFr tyrosine kinase inhibitors (e.g. erlotinib).
* Prior chemotherapy, radiotherapy or antibody therapy for gastric cancer or cancer of the gastro-oesophageal junction.
* Concomitant therapy with sorivudine or analogue compounds.
* Known previous or ongoing abuse of narcotic drug, other medication or alcohol.
* Significant cardiovascular disease including New York Heart Association (NYHA) grade II or greater congestive heart failure, peripheral arterial occlusive disease stage II or greater, symptomatic coronary heart disease, insufficiently treated arterial hypertension, unstable angina or myocardial infarction within 12 months before initiating study treatment or a history of ventricular arrhythmia.
* History or evidence upon physical examination of CNS disease unless adequately treated, seizure not controlled with standard medical therapy, or history of stroke.
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan.
* Pre-existing polyneuropathy grade >1 according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), except for loss of tendon reflex as the only symptom.
* Treatment for systemic infection within 14 days before initiating study treatment.
* Active inflammatory bowel disease, serious gastric ulceration or other bowel disease causing chronic diarrhoea (defined as > 4 loose stools per day).
* Suspected or known dihydropyrimidine dehydrogenase deficiency (DPD).
* Thrombosis or severe bleeding within six months prior to entry into the study (except for bleeding of the tumour before its surgical resection), evidence of bleeding diathesis or coagulopathy, or current or recent (within 10 days prior to initiation of study treatment) use of full-dose oral or parenteral anticoagulants for therapeutic purposes.
* History of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results.
* Known positive test for human immunodeficiency virus infection, hepatitis C virus or chronic active hepatitis B infection.
* Known allergy to the investigational product, to any of its excipients, to monoclonal antibodies, or to any of the components of the chemotherapy regimen.
* Any co-morbid disease that would increase risk of toxicity.
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures.
* Any investigational agent or participation in another clinical trial within 30 days prior to randomisation.
* Must not have had a major surgical procedure within 28 days of randomisation.
* Subject who is pregnant or breast feeding.
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions (intrauterine contraceptive device, contraceptive implants, injectables (hormonal depot), transdermal hormonal contraception (contraceptive patch), sexual abstinence or vasectomised partner) during the course of the study and for six months after the last study drug administration for women and men. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-child-bearing potential.
* Subject unwilling or unable to comply with study requirements.
* Hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Frequency of pT3/T4 categories after surgery | after 9 weeks treatment

SECONDARY OUTCOMES:
Frequencies of pN2/N3 categories after surgery | After 9 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: M. Stahl, Prof. Dr. med., Principal Investigator — Klinken Essen-Mitte Evang. Huyssens-Stiftung
Locations (1):
- AIO-Studien gGmbH, Berlin, Germany

REFERENCES:
- [Background] Becker K, Mueller JD, Schulmacher C, Ott K, Fink U, Busch R, Bottcher K, Siewert JR, Hofler H. Histomorphology and grading of regression in gastric carcinoma treated with neoadjuvant chemotherapy. Cancer. 2003 Oct 1;98(7):1521-30. doi: 10.1002/cncr.11660. PMID 14508841
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Background] Garcia I, del Casar JM, Corte MD, Allende MT, Garcia-Muniz JL, Vizoso F. Epidermal growth factor receptor and c-erbB-2 contents in unresectable (UICC R1 or R2) gastric cancer. Int J Biol Markers. 2003 Jul-Sep;18(3):200-6. doi: 10.1177/172460080301800308. PMID 14535591
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Derived] Stahl M, Maderer A, Lordick F, Mihaljevic AL, Kanzler S, Hoehler T, Thuss-Patience P, Monig S, Kunzmann V, Schroll S, Sandermann A, Tannapfel A, Meyer HJ, Schuhmacher C, Wilke H, Moehler M; Arbeitsgemeinschaft Internistische Onkologie (AIO) Oesophageal and Gastric Cancer Working Group and the Chirurgische Arbeitsgemeinschaft Onkologie (CAOGI/DGAV) of the German Cancer Society. Perioperative chemotherapy with or without epidermal growth factor receptor blockade in unselected patients with locally advanced oesophagogastric adenocarcinoma: Randomized phase II study with advanced biomarker program of the German Cancer Society (AIO/CAO STO-0801). Eur J Cancer. 2018 Apr;93:119-126. doi: 10.1016/j.ejca.2018.01.079. Epub 2018 Mar 20. PMID 29501977
- See also: Arbeitsgemeinschaft der internistischen Onkologie — http://www.aio-portal.de